CLINICAL TRIAL: NCT04650633
Title: A Phase II,Open-label Trial to Investigate the Efficacy and Safety of SHR-1701 in Patients With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: SHR-1701 in Patients With Recurrent/Metastatic Scchn
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-II-208
Record Dates: First submitted 2020-11-25; First posted 2020-12-02 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2020-11

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: SHR-1701; Phase II
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — SHR-1701

STUDY DESIGN:
Intervention Model Description: 2 cohorts
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1701 (Experimental): R/M SCCHN subjects failure after 1 lines of platinum based chemotherapy or after anti PD-1/PD-L1 antibody therapy.
  Interventions: Drug: SHR-1701

INTERVENTIONS:
Drug: SHR-1701 — Subjects will receive an intravenous infusion of SHR-1701 until confirmed progression, unaccepted toxicity, or any criterion for withdrawal from the trial.

SUMMARY:
This is an open label, single-arm, multi-center, phase II study of SHR-1701 in patients with recurrent/metastatic SCCHN

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Recurrent/Metastatic SCCHN,not include NPC
2. Subjects failure after 1 lines of platinum based chemotherapy or failure from anti-PD-1/PD-L1 antibody therapy.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at trial entry.
4. Disease must be measurable with at least 1 uni dimensional measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
5. Adequate hematological, hepatic and renal function as defined in the protocol Other protocol-defined inclusion criteria could apply.

Exclusion Criteria:

1. Prior therapy with an anti-PD1, anti-PD-L1, anti-CTLA-4 or a TGFb inhibitor.
2. Anticancer treatment within 28 days before the first dose of study drug.
3. Major surgery within 28 days before start of trial treatment.
4. Systemic therapy with immunosuppressive agents within 7 days prior to the first dose of study drug; or use any investigational drug within 28 days before the start of trial treatment.
5. With any active autoimmune disease or history of autoimmune disease.
6. History of immunodeficiency including seropositive for human immunodeficiency virus (HIV), or other acquired or congenital immunedeficient disease, or any active systemic viral infection requiring therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 | up to 2 years
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: at least 30% decrease in the sum of diameters of target lesions) per RECIST 1.1.

SECONDARY OUTCOMES:
DOR | 24 months
  Duration of response
DCR | 24 months
  Disease Control Rate
PFS | 24 months
  Progression free survival
OS | 24 months
  Overall Survival
AEs | 24 months
  Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Tumor Hospital of the Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided